CLINICAL TRIAL: NCT03618303
Title: Combined Positron Emission Tomography and Magnetic Resonance Imaging of Coronary Atherothrombosis
Brief Title: PET-MR Imaging of Coronary Atherothrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AC17091
Record Dates: First submitted 2018-07-31; First posted 2018-08-07 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Heart Diseases, Ischemic
MeSH Terms: conditions — Myocardial Ischemia | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): All patients will undergo the same intervention of having a PET-MRI scan and optical coherence tomography.
  Interventions: Diagnostic Test: PET-MRI scan

INTERVENTIONS:
Diagnostic Test: PET-MRI scan — Patients will undergo combined Positron Emission Tomography and Magnetic Resonance Imaging prior to a planned invasive angiogram (performed as standard of care). During the angiogram procedure, an additional imaging test (optical coherence tomography) will be performed.
  Other Names: Optical Coherence Tomography

SUMMARY:
Heart attacks remain a common cause of death throughout the world. The most common initiating event is the formation of a blood clot within the coronary arteries occluding blood supply to the heart. However, we know that thrombus often occurs within the coronary arteries without causing any symptoms, and may be found in patients with stable angina. We wish to investigate whether blood clots within the coronary arteries can be detected in patients who have had a heart attack and in patients with stable angina using combined positron emission tomography and magnetic resonance (PET-MR) imaging. If possible, this may provide a safe and noninvasive means of identifying patients at higher risk of heart attacks.

The study will be conducted in Edinburgh Heart Centre and a total of 40 participants will be recruited from the cardiology wards, outpatient clinics and day case unit. Participants will be asked to undergo a single PET-MRI scan in addition to invasive angiography as part of standard care (non-research procedure). During the invasive angiogram procedure, an additional imaging test may be performed called Optical Coherence Tomography to provide images from within the heart blood vessels.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed coronary artery disease undergoing elective invasive angiography OR
* Admitted with acute coronary syndrome diagnosed by two of the following criteria 1) Elevation of cardiac biomarkers (High sensitivity cardiac troponin I greater than 34 ng/l in men and 16ng/l in women) 2) Symptoms of myocardial ischaemia 3) ECG changes indicative of acute ischaemia

Exclusion Criteria:

* Contraindication or inability to undergo MRI scanning
* Renal failure (estimated glomerular filtration rate less than 30mL/min
* Undergoing Primary PCI
* Ongoing myocardial ischaemia or dynamic ECG changes
* Inability to provide informed consent
* Known allergy to gadolinium based contrast
* Women who are pregnant, breastfeeding or of child-bearing potential

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-03-24 (Actual); Study Completion 2020-03-24 (Actual)

PRIMARY OUTCOMES:
Plaque-to-myocardial ratio of culprit plaques on T1-weighted imaging | Baseline
  The identification of high risk plaques on T1-weighted MRI to determine whether coronary atherothrombosis can accurately be detected using non-invasive PET-MR imaging.

SECONDARY OUTCOMES:
The correlation between high risk plaques on PET-MR and culprit plaques on invasive angiography in patients with coronary artery disease. | Baseline
  The relationship between positive plaques identified on PET-MR by both T1-weighted MRI and 18F-NaF PET and culprit plaques on invasive angiography
The correlation between coronary plaque thrombosis (MRI), high-risk plaque (PET) and the presence of myocardial infarction on MRI (late enhancement). | Baseline
  The relationship between high risk plaque features on MRI and PET with evidence of myocardial infarction on MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Mhairi K Doris, MBChB, Principal Investigator — University of Edinburgh; David E Newby, PhD DM DSc, Study Chair — University of Edinburgh
Locations (1):
- Queen's Medical Research Institute, Edinburgh, Scotland, United Kingdom

REFERENCES:
- [Background] Xie Y, Kim YJ, Pang J, Kim JS, Yang Q, Wei J, Nguyen CT, Deng Z, Choi BW, Fan Z, Bairey Merz CN, Shah PK, Berman DS, Chang HJ, Li D. Coronary Atherosclerosis T1-Weighed Characterization With Integrated Anatomical Reference: Comparison With High-Risk Plaque Features Detected by Invasive Coronary Imaging. JACC Cardiovasc Imaging. 2017 Jun;10(6):637-648. doi: 10.1016/j.jcmg.2016.06.014. Epub 2016 Oct 12. PMID 27743950
- [Background] Noguchi T, Kawasaki T, Tanaka A, Yasuda S, Goto Y, Ishihara M, Nishimura K, Miyamoto Y, Node K, Koga N. High-intensity signals in coronary plaques on noncontrast T1-weighted magnetic resonance imaging as a novel determinant of coronary events. J Am Coll Cardiol. 2014 Mar 18;63(10):989-99. doi: 10.1016/j.jacc.2013.11.034. Epub 2013 Dec 15. PMID 24345595
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999
- [Background] Matsumoto K, Ehara S, Hasegawa T, Sakaguchi M, Otsuka K, Yoshikawa J, Shimada K. Localization of Coronary High-Intensity Signals on T1-Weighted MR Imaging: Relation to Plaque Morphology and Clinical Severity of Angina Pectoris. JACC Cardiovasc Imaging. 2015 Oct;8(10):1143-1152. doi: 10.1016/j.jcmg.2015.06.013. Epub 2015 Sep 9. PMID 26363839